CLINICAL TRIAL: NCT02614443
Title: Effectiveness and Acceptability of Internet-delivered Treatment for Depression, Anxiety and Stress in University Students: Protocol for an Open Feasibility Trial
Brief Title: Effectiveness and Acceptability of Internet-delivered Treatment for Depression, Anxiety and Stress
Acronym: EAITDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silver Cloud Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAITDAS
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Depression; Anxiety; Stress
Keywords: Depression; Anxiety; Stress; Online interventions; University students; CBT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Depression Condition (Experimental): Participants in this group will be offered the Space from Depression programme to be completed over an 8 week period. The programme is delivered through the online SilverCloud platform.
  Interventions: Other: Space from Depression
- Anxiety Condition (Experimental): Participants in this group will be offered the Space from Anxiety programme to be completed over an 8 week period. The programme is delivered through the online SilverCloud platform.
  Interventions: Other: Space from Anxiety
- Stress Condition (Experimental): Participants in this group will be offered the Space from Stress programme to be completed over an 8 week period. The programme is delivered through the online SilverCloud platform.
  Interventions: Other: Space from Stress

INTERVENTIONS:
Other: Space from Depression — Delivered through the online SilverCloud platform, the program for the treatment of depression employs several innovative engagement strategies for improving the user experience. These are divided into several categories: personal, interactive, supportive, and social.
  Arms: Depression Condition
Other: Space from Anxiety — Delivered through the online SilverCloud platform, the program for the treatment of anxiety employs several innovative engagement strategies for improving the user experience. These are divided into several categories: personal, interactive, supportive, and social.
  Arms: Anxiety Condition
Other: Space from Stress — Delivered through the online SilverCloud platform, the program for the treatment of stress employs several innovative engagement strategies for improving the user experience. These are divided into several categories: personal, interactive, supportive, and social.
  Arms: Stress Condition

SUMMARY:
The aims of this study are to test the effectiveness and acceptability of internet-delivered treatment for depression, anxiety and stress in university students. These data will inform the methods for a future randomized controlled trial.

The trial will establish an initial estimate of the effectiveness of these online interventions for students in terms of within-group effect sizes associated with changes in depression, anxiety and stress from pre to post-intervention and follow-up. These data will be used to estimate the sample size for a future trial to ensure that the study is sufficiently powered. A conservative estimate using the 90% upper confidence limit will be used to inform the sample size calculation of the definitive RCT.

Acceptability of the intervention to participants will be assessed using data on usage and engagement with the intervention (e.g. percentage of participants completing each module, average number of log ins, average time spent per session and total time spent on the program). These data are acquired through the online SilverCloud system. Satisfaction with will be assessed through the use of a post-intervention questionnaire on satisfaction with accessing and using an online delivery format for treatment.

DETAILED DESCRIPTION:
Depression, anxiety and stress are among the primary causes of disease rates worldwide and are the most prevalent mental health problems in the U.S. Each is associated with significant economic, personal, intrapersonal and societal losses including lower quality of life and increased mortality.

Depression, Anxiety and Stress in Students:

Depression and anxiety are also the most prevalent mental health problems among the student population. In the 2010 American College Health Survey, 48% of college and university students reported feeling overwhelming anxiety at least once in the previous year. Thirty-one percent reported feeling so depressed it was difficult to function at least once in the previous 12 months. More recently, University counseling and mental health services have reported an increase in the number of clients seeking services and in yearly visits.

The college years can be a highly stressful time in students' lives. This is particularly true of the period of transition to college as students are learning to cope with increased academic pressures. Students are at a developmental stage when newfound stressors can promote the onset of mental health difficulties. In addition to academic stress, international students can experience significant sociocultural adjustment demands.

Young adults between 17 and 25 years of age are reported to be at greater risk of developing a serious mental illness than individuals in other age groups. Although early diagnosis of mental disorders can be difficult, delayed diagnosis can often lead to treatment resistance and poorer longer-term outcomes. In addition, underachievement or failure at this point in life can cause long-term setbacks to individuals' self-esteem and future progress.

Treating Depression, Anxiety and Stress:

Depression, anxiety and stress disorders can each be treated effectively using medications; however, after completing a course of this type of treatment the chances of relapse are high, and equally successful psychological therapies are often preferred. Of these, cognitive-behavior therapy (CBT) is the most widely researched and CBT is recognized as the leading choice of treatment for depression and anxiety in terms of post-treatment improvements, maintaining progress, and preventing relapse. CBT also is effective for stress management. CBT is comprised of a variety of cognitive and behavioral approaches, each concerned with changing distressing thoughts and beliefs. Treatment is often comprised of self-monitoring and thought recording, behavioral activation, cognitive restructuring, and exposure.

Access to Treatment:

On a global scale, a significant number of individuals in need of treatment receive no medical diagnosis nor do they seek treatment. The worldwide treatment gap between those needing treatment for depression compared to those receiving treatment has been estimated at 56%; the gap in treatment for anxiety disorders has been estimated at 46%. Several factors prevent people from accessing treatment, such as waiting lists, lack of motivation, negative attitudes about treatment, and costs. Of those willing to seek treatment, many encounter a lack of trained professionals or are placed on a waiting list. Although students can often obtain mental health services on campus, many campuses have limited services or have wait lists for services because of the high demand. A survey of U.S. students with mental health problems revealed that common barriers to seeking services, even if they were available, were stigma, lack of time/accessibility, and wait lists. Internet-delivered interventions are one way to address these issues.

Internet-Delivered CBT (iCBT):

Internet-delivered CBT programs are specially designed for the treatment of specific disorders, and can be either clinician-guided or self-administered. When such interventions are used in the UK, 6-8 sessions is the recommended length of treatment. Many studies provide support for the utility and effectiveness of internet-delivered treatments for depression, anxiety and stress . Those with the additional feature of human support tend to produce greater results.

Several studies also have assessed the efficacy of online interventions for depression, stress, and anxiety for college students. Recent reviews of these studies have found evidence for the efficacy of these online interventions. However, most of these studies do not assess the efficacy of the interventions in the context of existing service delivery systems. Rather, many are RCTs assessing efficacy in convenience samples of students (e.g., Psychology majors). The current trial seeks to investigate the effectiveness and acceptability of internet-delivered interventions among university students seeking services and the procedures needed to incorporate these interventions into mental health delivery in U.S. universities. Additionally, it hopes to support and extend existing empirical evidence for SilverCloud programs.

University of Minnesota:

The University of Minnesota-Twin Cities is a public research university located in Minneapolis and St. Paul, Minnesota established in 1851. It is the oldest and largest campus within the University of Minnesota system and has the sixth-largest main campus student body in the United States, with 57,600 students. The university is organized into 19 colleges and schools.

Participants will be recruited through three units at the University of Minnesota-Twin Cities. The first is Student Counseling Services (SCS) which provides free short-term counseling to undergraduate and graduate students. The second is Boynton Mental Health Clinic (BMHC) which also provides short term psychological services to full-time students at the University of Minnesota. Unlike SCS, BMHC also has psychiatrists on staff and is affiliated with the university health service. Finally, the investigators will recruit participants through the International Student and Scholar Services (ISSS) office which provides counseling to foreign national students on campus.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age. Participants must have self-reported mild to severe symptoms of depression (5-27+) according to PHQ-9, self-reported mild to severe symptoms of anxiety (5-21+) according to GAD-7, or self-reported mild to severe symptoms of stress (15-34+) according to the stress sub-scale of DASS-21.

Exclusion Criteria:

* Students who currently are in face-to-face therapy at UCCS or BHS will be excluded. Students who score in the "red zone" in terms of risk of self-harm on the screening questions routinely used at UCCS will not be referred to the study. Students who score greater than 0 on the PHQ-9 self-harm item during the initial screening phase will be automatically directed to be further evaluated and alerted that a counselor will try to reach them. Based on this further evaluation, they may be recommended to seek help from their health/counseling service and may/may not be eligible to participate in the study. They will be telephoned within 1 working day and contacted by email if they cannot be reached by phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Stress sub-scale of Depression Anxiety and Stress Scale-21 (DASS-21) | Baseline, postintervention at 8 weeks and 3 month follow-up
  Composed of 7-item sub-scale measuring symptoms of stress.
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, postintervention at 8 weeks and 3 month follow-up
  A self-report measure of depression that has been widely used in screening, primary care, and research.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, postintervention at 8 weeks and 3 month follow-up
  Comprises 7 items measuring symptoms and severity of GAD based on the DSM-IV diagnostic criteria for GAD.

OTHER OUTCOMES:
Change in The Satisfaction with Treatment (SAT) Questionnaire | Postintervention at 8 weeks and 3 month follow-up
  Satisfaction measure containing two qualitative questions asking participants to describe what they most liked and least liked about the online treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — SilverCloud Health; Patricia Frazier, PhD, Principal Investigator — University of Minnesota; Stefan G. Hofmann, PhD, Principal Investigator — Department of Psychological and Brain Sciences, Boston University; Deborah Beidel, PhD, Principal Investigator — UCF RESTORES, Department of Psychology, University of Central Florida; Patrick A. Palmieri, PhD, Principal Investigator — Center for the Treatment and Study of Traumatic Stress, Summa Health System, Akron, Ohio; Jacqueline Mooney, MA, Principal Investigator — SilverCloud Health; Christopher Bonner, MSc, Principal Investigator — SilverCloud Health
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kessler RC, Aguilar-Gaxiola S, Alonso J, Chatterji S, Lee S, Ormel J, Ustun TB, Wang PS. The global burden of mental disorders: an update from the WHO World Mental Health (WMH) surveys. Epidemiol Psichiatr Soc. 2009 Jan-Mar;18(1):23-33. doi: 10.1017/s1121189x00001421. PMID 19378696
- [Background] Cuijpers P, Smit F, Oostenbrink J, de Graaf R, Ten Have M, Beekman A. Economic costs of minor depression: a population-based study. Acta Psychiatr Scand. 2007 Mar;115(3):229-36. doi: 10.1111/j.1600-0447.2006.00851.x. PMID 17302623
- [Background] Rapaport MH, Clary C, Fayyad R, Endicott J. Quality-of-life impairment in depressive and anxiety disorders. Am J Psychiatry. 2005 Jun;162(6):1171-8. doi: 10.1176/appi.ajp.162.6.1171. PMID 15930066
- [Background] Richards D. Prevalence and clinical course of depression: a review. Clin Psychol Rev. 2011 Nov;31(7):1117-25. doi: 10.1016/j.cpr.2011.07.004. Epub 2011 Jul 23. PMID 21820991
- [Background] Day V, McGrath PJ, Wojtowicz M. Internet-based guided self-help for university students with anxiety, depression and stress: a randomized controlled clinical trial. Behav Res Ther. 2013 Jul;51(7):344-51. doi: 10.1016/j.brat.2013.03.003. Epub 2013 Mar 28. PMID 23639300
- [Background] Adlaf EM, Gliksman L, Demers A, Newton-Taylor B. The prevalence of elevated psychological distress among Canadian undergraduates: findings from the 1998 Canadian Campus Survey. J Am Coll Health. 2001 Sep;50(2):67-72. doi: 10.1080/07448480109596009. PMID 11590985
- [Background] American College Health Association (2010). National college health assessment reference group executive summary. Hanover, MD: American College Health Association.
- [Background] Association for University and College Counseling Center Directors (2014). The Association for University and College Counseling Center Directors Annual Survey. Aurora, IL: Association for University and College Counseling Center Directors.
- [Background] Rutter M, Sroufe LA. Developmental psychopathology: concepts and challenges. Dev Psychopathol. 2000 Summer;12(3):265-96. doi: 10.1017/s0954579400003023. PMID 11014739
- [Background] Dyson R, Renk K. Freshmen adaptation to university life: depressive symptoms, stress, and coping. J Clin Psychol. 2006 Oct;62(10):1231-44. doi: 10.1002/jclp.20295. PMID 16810671
- [Background] Hirai R, Frazier P, Syed M. Psychological and sociocultural adjustment of first-year international students: Trajectories and predictors. J Couns Psychol. 2015 Jul;62(3):438-52. doi: 10.1037/cou0000085. Epub 2015 May 11. PMID 25961754
- [Background] Wang PS, Berglund PA, Olfson M, Kessler RC. Delays in initial treatment contact after first onset of a mental disorder. Health Serv Res. 2004 Apr;39(2):393-415. doi: 10.1111/j.1475-6773.2004.00234.x. PMID 15032961
- [Background] Johnson EM, Coles ME. Failure and delay in treatment-seeking across anxiety disorders. Community Ment Health J. 2013 Dec;49(6):668-74. doi: 10.1007/s10597-012-9543-9. Epub 2012 Sep 29. PMID 23054147
- [Background] Cuijpers P, Sijbrandij M, Koole SL, Andersson G, Beekman AT, Reynolds CF 3rd. Adding psychotherapy to antidepressant medication in depression and anxiety disorders: a meta-analysis. World Psychiatry. 2014 Feb;13(1):56-67. doi: 10.1002/wps.20089. PMID 24497254
- [Background] Richardson KM, Rothstein HR. Effects of occupational stress management intervention programs: a meta-analysis. J Occup Health Psychol. 2008 Jan;13(1):69-93. doi: 10.1037/1076-8998.13.1.69. PMID 18211170
- [Background] Donohue, E. O., & Fisher, J. E. (Eds.). (2012). Cosgitive Behavior Therapy: Core principles and practice. Hoboken, New Jersey: John Wiley & Sons.
- [Background] Alegria, M., Kessler, R. C., Bijl, R., Lin, E., Heeringa, S. G., Takeuchi, D. T., et al. (2000). Comparing mental health service use data across countries. In: Andrews G, editor. Unmet need in mental health service delivery. Cambridge: Cambridge University Press; p. 97-118
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Mohr DC, Ho J, Duffecy J, Baron KG, Lehman KA, Jin L, Reifler D. Perceived barriers to psychological treatments and their relationship to depression. J Clin Psychol. 2010 Apr;66(4):394-409. doi: 10.1002/jclp.20659. PMID 20127795
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Richards, D., & Timulak, L. (2012). Satisfaction with therapist-delivered vs. self-administered online cognitive behavioural treatments for depression symptoms in college students. British Journal of Guidance & Counselling, 41(2), 193-207. doi: 10.1080/03069885.2012.726347
- [Background] Richards, D., & Timulak, L. (2012). Client-identified helpful and hindering events in therapist delivered vs. self-administered online cognitive-behavioural treatments for depression in college students. Counselling Psychology Quarterly, 25, 251-262.
- Available data/document: Study Protocol: 10.1186/s40814-016-0068-9 — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-016-0068-9